CLINICAL TRIAL: NCT03003208
Title: Pulmonary Rehabilitation and Cardiovascular Risk in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16/0446
Record Dates: First submitted 2016-12-15; First posted 2016-12-26 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary rehabilitation (Other)
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — An exercise and education program

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common smoking-related lung disease. Patients with COPD are at increased risk of developing cardiovascular disease such as heart attacks and strokes. A simple measurement called arterial stiffness is a good assessment of how likely people are to have cardiovascular disease, both in healthy populations and those with COPD. Aortic Pulse wave velocity (aPWV) measures arterial stiffness,

Pulmonary Rehabilitation (PR) - a 6 week supervised group exercise and education class - is an effective intervention in COPD to reduce symptoms, improve exercise performance and prevent exacerbations. However, the effect of PR on cardiovascular risk in COPD is controversial as two small positive studies suggested benefit and one larger study did not.

Investigators have recently shown that cardiovascular risk is higher in those COPD patients who get the most infections (exacerbations). PR is an effective intervention for preventing COPD exacerbations. Logically, the exercise component would be expected to reduce cardiovascular risk too.

Investigators want to identify which patients with COPD get cardiovascular benefit from a PR programme and why others do not. Investigators propose to measure aPWV before and after PR. Investigators will then classify participants as responders or non-responders defined as the presence or absence of a significant improvement in aPWV. Investigators will be collecting demographic and clinical information including daily physical activity level and how effective the PR has been to enable the investigators to identify the characteristics of patients who do, and do not achieve cardiovascular risk reduction in response to PR in COPD. This will inform on better design of PR programmes for people living with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with COPD. The patient must be referred to PR from his/her physician with spirometry results confirming that he/she has chronic obstructive pulmonary disease (defined as post-bronchodilator FEV1/VC <0.70 and a compatible exposure history).
* Ability to exercise.

Exclusion Criteria:

* Neuromuscular diagnosis.
* Patient involved in any ongoing drug intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
arterial stiffness | 6 weeks
  aortic pulse wave velocity

SECONDARY OUTCOMES:
Exercise capacity | 6 weeks
  Incremental Shuttle Walk Test (ISWT)
Physical activity level | 6 weeks
  steps counter pedometer
Change in dyspnea | 6 weeks
  Medical Research Council (MRC) dyspnoea scale
patient quality of life | 6 weeks
  COPD (CAT) assessment test

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free Hospital NHS, London, NW3 2PF, United Kingdom

REFERENCES:
- [Derived] Aldabayan YS, Ridsdale HA, Alrajeh AM, Aldhahir AM, Lemson A, Alqahtani JS, Brown JS, Hurst JR. Pulmonary rehabilitation, physical activity and aortic stiffness in COPD. Respir Res. 2019 Jul 24;20(1):166. doi: 10.1186/s12931-019-1135-6. PMID 31340825